CLINICAL TRIAL: NCT01327859
Title: A 52-week, Multicentre Open Label Extension Study of the Safety Tolerability and Efficacy of Donepezil (Aricept) in Parkinson's Disease (PD) Patients With Dementia
Brief Title: Safety, Tolerability, and Efficacy of Donepezil (Aricept) in Parkinson' s Disease (PD) Patients With Dementia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Margaret Moline, PhD, Eisai Inc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2020-E044-318; 2004-003355-39 (EudraCT Number)
Record Dates: First submitted 2011-03-30; First posted 2011-04-04 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Parkinson's Disease; Dementia
MeSH Terms: conditions — Parkinson Disease; Dementia

ARMS (3):
- Prior Donepezil 5mg (Experimental)
  Interventions: Drug: Prior Donepezil 5mg
- Prior Donepezil 10mg (Experimental)
  Interventions: Drug: Prior Donzepezil 10mg
- Prior Placebo (Placebo Comparator)
  Interventions: Drug: Prior Placebo

INTERVENTIONS:
Drug: Prior Donepezil 5mg — Received 5 mg donepezil once daily during the preceding double-blind study, E2020-G000-316. Received open-label 5 or 10 mg donepezil during the present study.
  Arms: Prior Donepezil 5mg
Drug: Prior Donzepezil 10mg — Received 10 mg donepezil once daily during the preceding double-blind study, E2020-G000-316 . Received open-label 5 or 10 mg donepezil during the present study.
  Arms: Prior Donepezil 10mg
Drug: Prior Placebo — Received placebo once daily during the preceding double-blind study, E2020-G000-316. Received open-label 5 or 10 mg donepezil during the present study.
  Arms: Prior Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of donepezil (Aricept) in Parkinson's Disease (PD) patients with dementia.

DETAILED DESCRIPTION:
Patients who complete all 24 weeks of the double-blind study E2020-E044-316 (NCT00165815) will be eligible for the open label extension study. Patients and caregiver/study partner will need to provide additional written informed consent to participate in the open label extension study. Safety and tolerability will be assessed after 4, 8 12, 24, 36 and 52 weeks. Cognition, Global Clinical Function, Activities of Daily Living, and Behaviour will be assessed after 24, and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age range: patients must be aged 40 or over
* Sex distribution: male and female
* PD according to UK Brain Bank criteria 40 with good response to levodopa as judged by investigator opinion.
* Women of child bearing potential must have demonstrated a negative serum beta human chorionic gonadotropin (B-HCG) at the screening visit for the double-blind study (E2020-E044-316)(NCT00165815) and a negative urine test result at the screening visit for the open label extension study, (E2020-E044-318)
* Completed all 24 treatment weeks of the double-blind study E2020-E044-316 (NCT00165815)and completed assessments.
* Outpatients, with a responsible and reliable caregiver/study partner
* Health: generally healthy and ambulatory or ambulatory-aided (i.e., walker or cane); vision (glasses, contact lenses permissible), hearing (hearing aid permissible) and speech sufficient for compliance with testing procedures; must be capable of swallowing the study medication.
* Written informed consent must be obtained from each patient and his/her caregiver/study partner prior to subjecting the patient or caregiver/study partner to any open label extension study related procedures.

Exclusion Criteria:

* Pregnant or lactating, women.
* Women of childbearing potential unless:

  * surgically sterile or
  * must be practicing effective contraception (e.g. abstinence, IUD or barrier method plus hormonal method). These patients must be willing to remain on current form of contraception for the duration of the study, (post menopausal women must be amenorrheic for at least 12 months to be considered of non-child bearing potential).
* Patients with evidence of other psychiatric/neurological disorders, i.e., stroke, schizophrenia, seizure disorder, head injury with loss of consciousness (for at least 1 hour) within the past year, progressive supranuclear palsy, multisystem atrophy, or dementia complicated by other organic disease.
* Evidence of clinically significant, active gastrointestinal, renal, hepatic, endocrine or cardiovascular system disease. Evidence of second or third degree heart block. Patients with controlled hypertension (supine diastolic blood pressure (BP) < 95 mmHg), right bundle branch block (complete or partial) and pacemakers may be included in the study.
* Patients previously treated with centrally active acetylchlinesterase (AChE) inhibitors (e.g., physostigmine, tacrine, metrifonate, galantamine, rivastigmine, donepezil) except the medication in the Aricept double-blind study E2020-E044-316 (NCT00165815).
* Patients and/or caregivers/study partners who are unwilling or unable to fulfill the requirements of the study.
* Any condition which would make the patient or the caregiver/study partner, in the opinion of the investigator, unsuitable for the study.
* Patients with known hypersensitivity to AChE inhibitors.
* Patients who were non-compliant with the inclusion/exclusion criteria or with the study medication received in the preceding Aricept? double-blind study E2020-E044-316 (NCT00165815).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2003-03; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will primarily be assessed by recording of AEs | 52 weeks

SECONDARY OUTCOMES:
To assess the efficacy of open-label donepezil (5-10 mg/day) on cognition (ADAS) | 52 weeks
To assess the efficacy of open-label donepezil (5-10mg/day) on cognition(MMSE) | 52 weeks
To assess the efficacy of open-label donepezil (5-10 mg/day) on Global Function (CIBIC) | 52 weeks
To assess the efficacy of open-label donepezil (5-10 mg/day) on ADLs (DAD and Schwab and England scales) | 52 weeks
To assess the efficacy of open-label donepezil (5-10 mg/day) on behavior (NPI) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Harre, Study Director — Eisai Limited
Locations (1):
- Bath, Canterbury, United Kingdom